CLINICAL TRIAL: NCT05579873
Title: Double Plating Versus Single Plating Techniques in Midshaft Clavicle Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Kantonsspital Obwalden (Unknown); Spital Schwyz (Unknown); Stryker SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-00574
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-07

CONDITIONS: Clavicle Fracture
Keywords: Clavicle/injuries; Bone Plates; Non-Randomized Controlled Trials as Topic
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single plating technique: Choice of implant used for single plating left at descretion of treating surgeon.
  Interventions: Procedure: Clavicle plating
- Double plating technique: Double plating consist of one VariAx 2.0mm plate positioned on the superior aspect of the clavicula and a second VariAx 2.4mm or 2.7 mm on the anterior side. Use of this implant will be according to the device's cleared indications of use.
  Interventions: Procedure: Clavicle plating

INTERVENTIONS:
Procedure: Clavicle plating — VariAx 2.0mm + 2.4 or 2.7mm vs any other single plate

SUMMARY:
The goal of this mutlicenter quasi-randomized observational cohort study is to compare single vs double plating in patients with a midshaft clavicle fracture. The main question it aims to answer is:

1. Does low profile double plating of midshaft clavicle fractures with one 2.0mm plate and a second 2.4 or 2.7 mm plate lead to a lower rate of re-intervention when compared to either single superior or single anterior plating?

DETAILED DESCRIPTION:
Clavicle fractures account for 2% to 5% of all fractures in adults, with a majority of patients being young and active. A gold standard for the treatment of clavicle fractures has yet to be established, but single plated surgical intervention is most widely used. In recent years a smaller double plating technique has been described as a possible solution to the high removal rates associated with single plating. In (orthopaedic) surgery however, randomized controlled trials (RCTs) are recognized for their limitations. Although RCTs are considered the gold standard for testing the efficacy of new interventions, randomisation and blinding can be challenging. Simultaneously, there is an inclination for the usage of RCTs in clinical protocols, frequently based on the credo that it is the only valid method of comparing treatments. A natural experiment (NE), or quasi-experiments, in which groups are compared by nature of factors outside the control of the investigator (i.e. different surgical techniques between centres), offers a possible solution for methodological quality control. This study aims to increase the knowledge on surgical outcomes for single vs double plating in midshaft clavicle fractures following a natural experiment design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Primary mid-shaft clavicula fracture defined as the middle third of the clavicle (Robinson Type II or AO 15.2)
* Patients that are eligible for operative treatment of clavicle fractures.

Generally accepted indications include:

* Displacement of one or more shaft width
* Shortening of more than 1cm in length
* High demand patients (physical activity)

Exclusion Criteria:

* Delayed presentation (> 14 days)
* Initial operative treatment at non-participating hospitals
* Open fractures
* Pathological fractures
* Re-fractures of clavicle
* Concomitant ipsilateral injury of upper extremity (including but not limited to shoulder, scapula, and ribs)
* Cognitive impairment or language barrier precluding answering questionnaires
* Unable to complete follow-up (e.g. different residential area/tourists)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (>18 older) presenting at the emergency department (ED) or outpatient clinic with midshaft clavicle fractures.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of surgical re-interventions | 2 years follow-up
  Any type of re-intervention (i.e. plate removal, screw adjustment etc.)

SECONDARY OUTCOMES:
Number of surgical re-interventions | 1 year follow-up
  (including implant removal)
Fracture realted infections | 2 years follow-up
  According to metsemakers et al, 2018 (Metsemakers WJ, Morgenstern M, McNally et al., MHJ. Fracture-related infection: A consensus on definition from an international expert group. Injury. 2018 Mar;49(3):505-510. doi: 10.1016/j.injury.2017.08.040. Epub 2017 Aug 24. PMID: 28867644)
Symptomatic non union | 1 year follow-up
  defined as absence of radiological signs of healing (callus formation or fading of fracture lines) combined with pain at the fracture site at 12 months.
Asymptomatic non-union | 1 year follow-up
  defined as absence of radiological signs of healing (callus formation or fading of fracture lines) without any clinical symptoms.
Numbness below scar line | 1 year follow-up
  Tested postoperatively and at 12 months follow-up
Self-reported implant irritation/implant prominence | 1 year follow-up
  According to Hulsman et al, 2018 (17. Hulsmans M, van Heijl M, Houwert R, et al., Intramedullary nailing of displaced midshaft clavicle fractures using a TEN with end cap: issues encountered. Acta Orthop Belg. 2018 Dec;84(4):479-484. PMID: 30879453.)
Operative time | Baseline
Length of surgical incision | basline
  Length of surgical incision in cm
DASH score | baseline, 3- and 12-monts follow-up
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
EQ-5D | baseline (pre-injury), 3- and 12-months follow-up
  to monitor changes in self-reported health status through time in a given patient group
VAS pain score | 3- and 12-months follow-up
  Self-reported pain on a scale of 0 to 10.
VAS for patient satisfaction | 3- and 12-months follow-up
  Self-reported satisfaction on a scale of 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Frank Beeres, PhD/M.D., Principal Investigator — Chefarzt Chirurgie, speziell Unfallchirurgie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Meijden OA, Gaskill TR, Millett PJ. Treatment of clavicle fractures: current concepts review. J Shoulder Elbow Surg. 2012 Mar;21(3):423-9. doi: 10.1016/j.jse.2011.08.053. Epub 2011 Nov 6. PMID 22063756
- [Background] Robinson CM. Fractures of the clavicle in the adult. Epidemiology and classification. J Bone Joint Surg Br. 1998 May;80(3):476-84. doi: 10.1302/0301-620x.80b3.8079. PMID 9619941
- [Background] McKee RC, Whelan DB, Schemitsch EH, McKee MD. Operative versus nonoperative care of displaced midshaft clavicular fractures: a meta-analysis of randomized clinical trials. J Bone Joint Surg Am. 2012 Apr 18;94(8):675-84. doi: 10.2106/JBJS.J.01364. PMID 22419410
- [Background] Devji T, Kleinlugtenbelt Y, Evaniew N, Ristevski B, Khoudigian S, Bhandari M. Operative versus nonoperative interventions for common fractures of the clavicle: a meta-analysis of randomized controlled trials. CMAJ Open. 2015 Nov 10;3(4):E396-405. doi: 10.9778/cmajo.20140130. eCollection 2015 Oct-Dec. PMID 26770963
- [Background] Althausen PL, Shannon S, Lu M, O'Mara TJ, Bray TJ. Clinical and financial comparison of operative and nonoperative treatment of displaced clavicle fractures. J Shoulder Elbow Surg. 2013 May;22(5):608-11. doi: 10.1016/j.jse.2012.06.006. Epub 2012 Sep 7. PMID 22960145
- [Background] Chen MJ, DeBaun MR, Salazar BP, Lai C, Bishop JA, Gardner MJ. Safety and efficacy of using 2.4/2.4 mm and 2.0/2.4 mm dual mini-fragment plate combinations for fixation of displaced diaphyseal clavicle fractures. Injury. 2020 Mar;51(3):647-650. doi: 10.1016/j.injury.2020.01.014. Epub 2020 Jan 9. PMID 31948781
- [Background] Zhang F, Chen F, Qi Y, Qian Z, Ni S, Zhong Z, Zhang X, Li D, Yu B. Finite element analysis of dual small plate fixation and single plate fixation for treatment of midshaft clavicle fractures. J Orthop Surg Res. 2020 Apr 15;15(1):148. doi: 10.1186/s13018-020-01666-x. PMID 32295608
- [Background] Rompen IF, van de Wall BJM, van Heijl M, Bunter I, Diwersi N, Tillmann F, Migliorini F, Link BC, Knobe M, Babst R, Beeres FJP. Low profile dual plating for mid-shaft clavicle fractures: a meta-analysis and systematic review of observational studies. Eur J Trauma Emerg Surg. 2022 Aug;48(4):3063-3071. doi: 10.1007/s00068-021-01845-3. Epub 2022 Mar 2. PMID 35237845
- [Background] Metsemakers WJ, Morgenstern M, McNally MA, Moriarty TF, McFadyen I, Scarborough M, Athanasou NA, Ochsner PE, Kuehl R, Raschke M, Borens O, Xie Z, Velkes S, Hungerer S, Kates SL, Zalavras C, Giannoudis PV, Richards RG, Verhofstad MHJ. Fracture-related infection: A consensus on definition from an international expert group. Injury. 2018 Mar;49(3):505-510. doi: 10.1016/j.injury.2017.08.040. Epub 2017 Aug 24. PMID 28867644
- [Background] Hulsmans M, van Heijl M, Houwert R, Verleisdonk EJ, Frima H. Intramedullary nailing of displaced midshaft clavicle fractures using a TEN with end cap: issues encountered. Acta Orthop Belg. 2018 Dec;84(4):479-484. PMID 30879453
- [Background] Germann G, Harth A, Wind G, Demir E. [Standardisation and validation of the German version 2.0 of the Disability of Arm, Shoulder,Hand (DASH) questionnaire]. Unfallchirurg. 2003 Jan;106(1):13-9. doi: 10.1007/s00113-002-0456-x. German. PMID 12552388
- [Derived] Lecoultre Y, van de Wall BJM, Diwersi N, Pfarr SW, Galliker B, Babst R, Link BC, Beeres FJP. A natural experiment study: Low-profile double plating versus single plating techniques in midshaft clavicle fractures-Study protocol. PLoS One. 2023 Sep 8;18(9):e0291238. doi: 10.1371/journal.pone.0291238. eCollection 2023. PMID 37683048
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf